CLINICAL TRIAL: NCT02916537
Title: A Phase 1 Trial for Evaluation of the Safety, Pharmacokinetics, and [18F] Radiation Dosimetry of CTT1057, a Small Molecule Inhibitor of Prostate Specific Membrane Antigen (PSMA)
Brief Title: A Phase 1 Trial for Evaluation of the Safety, Pharmacokinetics, and [18F] Radiation Dosimetry of CTT1057
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Targeted Technology (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1057-101
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate specific membrane antigen; prostate neoplasms; metastatic prostate cancer; prostatic hyperplasia
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A: Pre-prostatectomy patients (Experimental): Patients with prostate cancer prior to radical prostatectomy (N = 5). Single IV dose (370 MBq, or 10 mCi). Combined PET/MR imaging (prostate + whole body) will be performed following tracer injection. Patients in cohort A will undergo radical prostatectomy (plus lymph node dissection) within 12 weeks following CTT1057 PET/MR.
  Interventions: Drug: CTT1057; Procedure: Prostatectomy
- Cohort B: Metastatic prostate cancer (Experimental): Patients with evidence of metastatic castration-resistant prostate cancer (N = 15).
  Single IV dose (370 MBq, or 10 mCi). Combined PET/MR imaging (prostate + whole body) will be performed following tracer injection. Patients in cohort B (metastatic prostate cancer) will have the option for metastatic tumor biopsy following CTT1057 PET imaging.
  Interventions: Drug: CTT1057

INTERVENTIONS:
Drug: CTT1057 — Single IV dose (370 MBq, or 10 mCi) of CTT1057 followed by combined PET/MR imaging (prostate + whole body).
Procedure: Prostatectomy — Radical prostatectomy with lymph node dissection
  Arms: Cohort A: Pre-prostatectomy patients

SUMMARY:
The purpose of this study is to test a novel diagnostic Positron Emission Tomography (PET) imaging agent for safety and biodistribution. The agent binds Prostate Specific Membrane Antigen (PSMA) and is designed to detect prostate tumors.

DETAILED DESCRIPTION:
The sponsor has developed a PET imaging agent, CTT1057, labeled with 18F, that is based on a small molecule core and targets an extracellular region of PSMA with high affinity. Although comparable to other inhibitors in terms of affinity for PSMA, this unique class of phosphoramidate agents are the only known irreversible PSMA inhibitors. Due to its irreversible binding to PSMA and rapid uptake by PSMA-expressing prostate cancer cells, accumulation at the cancer target is expected to be rapid, specific and sensitive.

Twenty patients will be enrolled in parallel in two cohorts:

* (Cohort A) Patients with prostate cancer prior to radical prostatectomy (N = 5).
* (Cohort B) Patients with evidence of metastatic castration-resistant prostate cancer (N = 15)

Participants receive a single intravenous (IV) dose (370 MBq, or 10 mCi) of CTT1057 in this first-in-human trial. Combined PET/MR imaging (prostate + whole body) will be performed following tracer injection. The 5 patients in the pre-prostatectomy cohort will comprise the dosimetry/pharmacokinetic (PK) cohort to establish organ dosimetry and PK profile. Patients in cohort A will undergo planned radical prostatectomy (plus lymph node dissection) within 12 weeks following CTT1057 PET/MR. Patients in cohort B (metastatic prostate cancer) will have the option for metastatic tumor biopsy following CTT1057 PET imaging.

The one-time nominal injected dose will be 370 MBq (10 mCi). Estimated mass dose is 20 µg of CTT1057. Dose will be in a volume of 3 - 5 mL, and will be injected intravenously as a bolus injection.

Vital signs, adverse event assessment, and 12 lead ECGs will be performed on day 1 before and after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male patients age ≥18 years old
* Histologically confirmed adenocarcinoma of the prostate
* Adequate organ function including:
* - Platelet count of > 50,000/mm3
* - Neutrophil count of > 1000/mm3
* - Serum Cr < 1.5 x ULN or estimated GFR > 60 ml/min based upon Cockroft-Gault equation
* - Proteinuria < 1 g/24 hours based upon 24 hour urine collection or spot urine protein/creatinine ratio
* - AST and ALT < 2.5 x ULN (< 5 x ULN in patients with known liver metastases)
* - Total bilirubin < 1.5 x ULN (< 3 x ULN in patients with known/suspected Gilbert's disease)
* ECOG performance status of 0 or 1
* Able to provide written informed consent and willing to comply with protocol requirements
* No contra-indication to MR including severe claustrophobia, incompatible aneurysm clips or cardiac pacemaker
* For men of childbearing potential, the use of effective contraceptive methods during the trial and within 6 months following radiotracer injection
* Cohort A only (N = 5 evaluable patients):- Planned radical prostatectomy within 12 weeks following protocol scan
* - No androgen deprivation, anti-androgen therapy, chemotherapy, or investigational systemic therapy prior to CTT1057 PET imaging
* Cohort B only:- Presence of at least three distinct metastatic lesions by standard imaging including whole body bone scan + cross-sectional imaging of the abdomen and pelvis obtained within 12 weeks prior to protocol scan
* - Castration-resistant disease as defined by PCWG2 criteria
* - Must remain on androgen deprivation therapy for duration of trial if no prior bilateral orchiectomy

Exclusion Criteria:

* Inadequate venous access per assessment of treating health care provider
* Receipt of radioisotope within 5 physical half lives prior to trial enrollment
* Prior treatment with alpha radiation therapy (Radium Ra 223 chloride; Xofigo™) during the previous 60 days
* Have a medical condition or other circumstances that, in the opinion of the investigator would significantly decrease the chances of obtaining reliable data, achieving the study objectives, or completing the trial.
* Histologic evidence of small cell prostate cancer or neuroendocrine differentiation in > 50% of biopsy tissue

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Adverse event frequency as graded by Common Toxicity Criteria version 4.03 | 7 days from time of injection

SECONDARY OUTCOMES:
Organ dosimetry/tissue uptake of CTT1057 as measured by PET/MR imaging of prostate cancer | Up to six hours from time of injection
Pharmacokinetic profile of CTT1057 as measured by radiotracer detection in blood samples | Up to four hours from time of injection
Level of CTT1057 uptake on PET/MR imaging of localized prostate cancer with PSMA protein expression by immunohistochemistry from subsequent radical prostatectomy specimens | 12 weeks
Optimal Standardized Uptake Value (SUV) ratio threshold on CTT1057 PET/MR for discriminating tumor pathology from primary prostate cancer tissue | 4 hours
Sensitivity and specificity of CTT1057 PET imaging on a lesion-by-lesion basis as compared with standard imaging in metastatic prostate cancer | 4 hours
Number of positive lesions on CTT1057 PET/MR in subjects with equivocal or negative conventional imaging scans | 4 hours
Location of positive lesions on CTT1057 PET/MR in subjects with equivocal or negative conventional imaging scans | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Langton-Webster, PhD, Study Chair — Cancer Targeted Technology
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided